CLINICAL TRIAL: NCT03242330
Title: Implant Survival in Two-piece Versus Single-piece Patient-specific Titanium Subperiosteal Implants in Atrophied Edentulous Mandibles: Randomized Clinical Trial
Brief Title: Two-piece Versus Single-piece Patient-specific Titanium Subperiosteal Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Ahmed Roshdy, Assistant lecturer, Department of Prosthodontics, Faculty of Oral and Dental Medicine, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cairo Uni
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Dental Implant
Keywords: Implant survival; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Dental Implantation, Subperiosteal

STUDY DESIGN:
Masking Description: After assignment to interventions, blinding of trial participants, care providers and outcome assessors is not applicable. Data analysts will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-piece subperiosteal implant (Experimental): The two-piece subperiosteal implant will be designed with an internal connection that will receive its prosthetic counterpart later in the second stage surgery, which will retain the final prosthesis in place. Two-piece constructions allow for undisturbed submerged healing, without being exposed to the oral environment, achieved by attaining primary closure over the inserted implant body.
  Interventions: Device: Subperiosteal implant
- Single-piece subperiosteal implant (Active Comparator): The single-piece subperiosteal implant will be designed in the from of a framework with protruding posts that will appear penetrating through the mucosa, and will later carry the overlying superstructure (prosthesis). Single-piece subperiosteal implants do not require a second stage surgery.
  Interventions: Device: Subperiosteal implant

INTERVENTIONS:
Device: Subperiosteal implant — Subperiosteal implants are placed and fitted 'onto' the jaw bone just right below the mucoperiosteum; where the post of the metal frame is in a protruding position through the mucosa holding the prosthesis that will be later fitted.

SUMMARY:
The objective of this trial is to find out if there is a difference between single-piece and two-piece titanium patient-specific mandibular subperiosteal implants in terms of implant survival, patient satisfaction, and soft tissue dehiscence. This is to enhance both surgical and prosthetic outcomes for the sake of improved implant longevity, soft tissue health and patient well-being.

DETAILED DESCRIPTION:
After obtaining a thorough medical and dental history and performing necessary laboratory investigations, the following steps will be undertaken:

Preoperative prosthetic preparation:

* For eligible patients who are already wearing upper and lower complete dentures: The dentures will be checked for adaptation, fit, stability and occlusion.
* For eligible patients who are not wearing upper and lower complete dentures:

Preliminary alginate impressions will be made using a perforated stock tray for both the maxillary and mandibular arches. Impressions are then poured into dental stone to obtain the diagnostic models. Occlusion blocks will be constructed over the diagnostic models, followed by bite registration, try-in and delivery of upper and lower complete dentures.

Afterwards, approved complete dentures will be duplicated using laboratory condensation silicone to construct a radiographic stent. The radiographic stent is prepared by using a ratio of 3:1 acrylic resin to barium sulphate mixture, and then the patient is sent for a Cone Beam Computed Tomography (CBCT) scan.

CBCT scanning and virtual design of the patient-specific implant (PSI):

The CBCT scan of the patients - in the form of DICOM files - will be imported into surgical planning software (Mimics 19, Materialise, Leuven, Belgium). A segmentation process will be accomplished by using the two dimensional CT cuts to define the image thresholds based on Hounsfield's units, excluding soft tissue and only highlighting hard tissue (bone). The maxilla/mandible region will be further isolated by cropping and/or region-growing functions to remove artifacts and select only the area of interest, followed by the 3D calculation of the selected regions. The 3D models will be exported in standard triangulation language (STL) format.

The STL files will then be imported into computer-aided design (CAD) software (3-matic) in order to create the design of the PSI. The subperiosteal part of the PSI will be drawn on the surface of the region planned to receive the PSI and then extruded to a thickness of 2.5mm. The PSIs will be meshed out with 2.5 mm holes to be compatible with 2.0 mm fixation screws. For the single-piece PSI, the abutments will be placed, guided by the opposing teeth and the radio-opaque dentures. As for the two-piece PSI, the same design will be repeated without the addition of the abutment posts.

Fabrication of the patient-specific implant (PSI):

The STL file of the final design will be sent for 3D printing via additive manufacturing using selective laser sintering (SLS) machine from medical titanium grade (Ti-6Al-4V) Extra Low Interstitials (ELI).

PSI surface treatment:

The PSI will be subjected to acid etching following a protocol proposed by Juodzbalys et al to attain micro roughness on the fitting surface of the implant. The PSIs will be etched with sulfuric acid (H2SO4) for 72 hours followed by Hydrochloric acid (HCl) for 30 hours. After removal from the acids PSIs will be washed in distilled water.

Cleaning and sterilization:

Implants will be cleaned in an ultrasonic bath of absolute ethyl alcohol solution at ambient temperature for 30 minutes to ensure the removal of any residues on the fitting surface of the implant. After being thoroughly cleaned, the PSIs will be wrapped and sterilized using a class B autoclave.

Surgical phase:

For both groups, under general anesthesia; a mucosal incision 3-5 mm crestal to the vestibule will be made in the anterior region similar to the genioplasty incision, followed by dissection over the orbicularis oris and mentalis muscle and incising down to bone using a scalpel blade #15c mounted on a Bard-Parker® surgical blade handle size 3, to expose the proposed implant site. The incision will be completed posteriorly after localization of the mental nerves. After bone exposure the implant will be installed in place and fixed with 2.0mm grade 5 titanium screws.

For two-piece PSIs, the framework will be designed with 3-4 mm endosseous projections at the anticipated area where the final abutments will be fastened, guided by the position of the teeth in the proposed prosthetic set-up. The endosseous projections will be designed in order to accommodate the height of the internal connection that will receive the final abutment in a second-stage surgery. Unlike single piece PSIs, bone-supported surgical guides will be designed to aid in the placement and seating of the two-piece PSIs corresponding to the preplanned osteotomy sites. The flap will be sutured in two layers; the muscle layer will be closed with 3/0 poliglecaprone resorbable suture material and the mucosa with 4/0 Polypropylene non-resorbable suture material.

Postoperative care and instructions:

The intra oral wounds will be evaluated for any signs of bleeding, hematoma, infection, wound dehiscence or PSI exposure after 48 hours, then weekly till the end of the first month. The following medications will be administered:

Long acting corticosteroids: Methylprednisolone Acetate 40 mg/ml intramuscular injection single dose immediate postoperative.

Anti-inflammatory analgesic: Ketorolac tromethamine 30 mg/amp/2mL intramuscular injection every 12 hours for the first 24 hours followed by diclofenac potassium 50 mg tablets (every 8 hours for 4 days) Oral antibiotic: Ampicillin/sulbactam 375 mg tablets (every 8 hours for 10 days) Strict oral hygiene measures in the form of regular use of chlorohexidine Gluconate 125 mg/100 mL antiseptic mouth wash (every 8 hours for two weeks).

Prosthetic phase:

The steps of fabrication of the final prosthesis will be initiated 3 months after implant placement for both groups. For the single-piece PSI group, a closed impression will be made. For the two-piece PSI group, final abutments will be fastened to the corresponding connection in the framework in a second stage surgery, followed by a final closed impression a week later. The final restoration will be constructed from a high impact polymer composite (HIPC) material via computer numerically controlled (CNC) milling. Occlusal adjustments will be performed followed by temporary cementation for two weeks until a final approval is obtained from the patient. Later, the prosthesis will be cemented using glass ionomer self-cured luting cement.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous male or female patients with atrophied mandibles between the ages of 50 to 75.
* Atrophic mandibular ridges in terms of width and height, impeding the possibility of placing a root form dental implant of at least 3mm in diameter and 8 mm in length.
* Completely edentulous patients (with the above mentioned criteria) who can't stand a soft-tissue supported mandibular denture.

Exclusion Criteria:

* Patients having a medical condition that absolutely contraindicates implant placement.
* Patients with uncontrolled diabetes, assessed by measuring glycosylated haemoglobin (HbA1c). Patients with an HbA1c level greater than 8 will be excluded.
* Potentially uncooperative patients who are not willing to go through the proposed interventions.
* Moderate-to-heavy daily smokers* (who report consuming at least 11 cigarettes/day).
* Patients who are satisfied with their soft-tissue supported mandibular denture.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 12 months (post-surgery)
  Implant survival will be assessed by evaluation of the following criteria:
  a) Persistent pain, and/or b) mobility and/or c) persistent exudate In case of presence of one or more of the previously mentioned criteria, implants will be regarded non-survived.
  Presence of persistent pain either spontaneous or during function Presence of clinically detected mobility Evidence of infection in the form of pus formation or persistent inflammatory fluid exudate

SECONDARY OUTCOMES:
Implant survival | 6 months (post-surgery)
  Implant survival will be assessed by evaluation of the following criteria:
  a) Persistent pain, and/or b) mobility and/or c) persistent exudate In case of presence of one or more of the previously mentioned criteria, implants will be regarded non-survived.
  Presence of persistent pain either spontaneous or during function Presence of clinically detected mobility Evidence of infection in the form of pus formation or persistent inflammatory fluid exudate
Implant survival | 3 months (post-surgery)
  Implant survival will be assessed by evaluation of the following criteria:
  a) Persistent pain, and/or b) mobility and/or c) persistent exudate In case of presence of one or more of the previously mentioned criteria, implants will be regarded non-survived.
  Presence of persistent pain either spontaneous or during function Presence of clinically detected mobility Evidence of infection in the form of pus formation or persistent inflammatory fluid exudate
Patient satisfaction | At 1,3,6 and 12 months (after loading of final prosthesis)
  Patient satisfaction is regarded an indicator of quality of healthcare. In this trial, the numerical rating scale (NRS) for patient satisfaction will be used, where patients will be asked to rate their satisfaction on the NRS (11-point ordinal scale) by selecting a whole number (0-10 integers), from 0 (completely dissatisfied) to 10 (completely satisfied). Higher scores portray higher satisfaction.
Soft tissue dehiscence | At 1,3,6 and 12 months (post-surgery)
  The investigators will subjectively assess this outcome through clinical examination of the oral tissues. It will be a binary outcome dichotomized to presence or absence of soft tissue breakdown based on the clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam A. Roshdy, Principal Investigator — Assistant lecturer, Department of Prosthodontics, Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sconzo J. The complete mandibular subperiosteal implant: an overview of its evolution. J Oral Implantol. 1998;24(1):14-5. doi: 10.1563/1548-1336(1998)242.0.CO;2. No abstract available. PMID 9759036
- [Background] Burns DR, Unger JW, Elswick RK Jr, Beck DA. Prospective clinical evaluation of mandibular implant overdentures: Part I--Retention, stability, and tissue response. J Prosthet Dent. 1995 Apr;73(4):354-63. doi: 10.1016/s0022-3913(05)80331-2. PMID 7783014
- [Background] Aras E, Sonmez M, Zora M, Basarir M, Kurtulmus H. The use of prefabricated titanium tissue abutments for the construction of a maxillary subperiosteal implant. J Oral Implantol. 2005;31(5):255-8. doi: 10.1563/1548-1336(2005)31[255:TUOPTT]2.0.CO;2. PMID 16265856
- [Background] OBWEGESER HL. Experiences with subperiosteal implants. Oral Surg Oral Med Oral Pathol. 1959 Jul;12(7):777-86. doi: 10.1016/0030-4220(59)90027-1. No abstract available. PMID 13674677
- [Background] The glossary of prosthodontic terms. J Prosthet Dent. 2005 Jul;94(1):10-92. doi: 10.1016/j.prosdent.2005.03.013. No abstract available. PMID 16080238
- [Background] Weiss CM, Reynolds T. A collective conference on the utilization of subperiosteal implants in implant dentistry. J Oral Implantol. 2000;26(2):127-8. doi: 10.1563/1548-1336(2000)262.0.CO;2. No abstract available. PMID 11831330
- [Background] Falomo OO, Hobkirk JA. A retrospective survey of patients treated with subperiosteal and endosseous implants. J Prosthet Dent. 1988 Nov;60(5):587-90. doi: 10.1016/0022-3913(88)90219-3. No abstract available. PMID 3058941
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Juodzbalys, G., M. Sapragoniene, and A. Wennerberg, New acid etched titanium dental implant surface. Stomatologija-Baltic Dental and Maxillofacial Journal, 2003. 5: p. 101-105.